CLINICAL TRIAL: NCT04037020
Title: Assessment of Dopaminergic Neurotransmission in Response to Tasting Chocolate (The Chocolate Study 2.0)
Brief Title: The Chocolate Study 2.0
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC218
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Normal Weight
MeSH Terms: interventions — Chocolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chocolate: Participants will be asked to taste commercially available chocolate varying in sugar, fat and percent cocoa.
  Interventions: Other: Chocolate

INTERVENTIONS:
Other: Chocolate — Participants will be asked to taste commercially available chocolate varying in sugar, fat and percent cocoa (extreme dark (90%), dark (70%), milk (38%), and white (0%)).

SUMMARY:
The purpose of this study is to test how the brain responds when enjoyable foods such as chocolate are consumed. The investigators know that eating certain types of foods can make an individual want to keep eating even when he or she is full. The chemical in the brain that causes this is called dopamine. The investigators can measure this response by looking at changes to how an individual's eye responds to light.

DETAILED DESCRIPTION:
The overall objective of this study is to determine dopamine (DA) neuromodulation (changes in b-wave amplitude as measured by electroretinography (ERG)) in response to consuming a highly reinforcing food (chocolate). The investigators hypothesize that orosensory stimulation with chocolates with increasing sugar content will increase the beta wave (b-wave) amplitude and the increase in the b-wave amplitude will correlate with score changes on the Psychophysical Effects Questionnaire (PEQ). This will be accomplished by testing different chocolates (extreme dark (90% cocoa), dark (70% cocoa), milk (38% cocoa), and white (0% cocoa)) on different days using 1.0 cd∙s/m2 flash luminance energy.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-24.9 kg/m2
* ability to understand and sign the consent form
* availability of transportation (i.e., participants must be able to provide their own transportation to the Grand Forks Human Nutrition Research Center)
* be free of any major illness/disease

Exclusion Criteria:

* food allergies
* participation in a weight loss diet/exercise program
* pregnancy
* lactation
* metabolic illness/disease (diabetes, renal failure, thyroid illness, hypertension)
* eye illness/disease (narrow angle glaucoma, macular degeneration, retinal detachment, cataracts)
* psychiatric, neurological or eating disorders (schizophrenia, depression, Parkinson's Disease, Huntington's Disease, cerebral palsy, stroke, epilepsy, anorexia nervosa or bulimia nervosa)
* taking any type of prescription medication with the exception of oral contraceptives and antihyperlipidemia agents

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Retinal dopamine response to oral stimuli | 30 minutes
  Electroretinograph b-wave amplitude will increase in response to increases in the amount of sugar in the chocolate.

SECONDARY OUTCOMES:
Correlation between b-wave amplitude and PEQ scores | 30 minutes
  The change in b-wave amplitude will positively correlate to Psychophysical Effects Questionnaire (PEQ) score changes.
Correlation between b-wave amplitude and habitual dietary intake | 30 minutes
  A preference for dark chocolate and/or a greater habitual fat intake will positively correlate with the retinal dopamine-mediated response to the dark chocolates (90% and 70% cocoa) and a preference for milk chocolate and/or a greater habitual added sugar will positively correlate with the retinal dopamine-mediated response to the milk and white chocolates. Higher amounts of artificial sweetener intake will will positively correlate with the retinal dopamine-mediated response to the milk and white chocolates. Greater habitual chocolate intake will positively correlate to changes in b-wave amplitude.

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT04037020/ICF_000.pdf